CLINICAL TRIAL: NCT03208699
Title: Screening and Diagnosis Help of Eating Disorders
Brief Title: EXPert System, ALImentary
Acronym: EXPALI
Status: Completed | Type: Observational
Sponsor: Marie-Pierre TAVOLACCI (Other)
Responsible Party: Sponsor-Investigator, Marie-Pierre TAVOLACCI, Docteur, University Hospital, Rouen
Organization: University Hospital, Rouen (Other)
Other Study IDs: 2017/124/OB
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Eating Disorder Symptom
Keywords: anorexia; bulimia
MeSH Terms: conditions — Anorexia; Bulimia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eating disorders (ED) are often undetected in the general population resulting in delayed treatment. The SCOFF questionnaire has been validated for eating disorders screening in primary care, but does not identify the type of eating disorder.

Objective: Investigators evaluated the performance of a clinical algorithm (ExpaliTM) combining answers to SCOFF questionnaire with Body Mass Index (BMI) to identify four Broad Categories of ED derived from DSM-5.

Design: Clinical algorithm (ExpaliTM) was developped from 104 combinations of BMI levels and answers to five SCOFF questions. Two senior ED specialists allocated each combination to one of the four Broad Categories of ED (DSM-5 diagnostics): restrictive disorder (anorexia nervosa typical, atypical and restrictive food intake disorders), bulimic disorder (typical and with low frequency or duration), hyperphagic disorder (binge eating disorders typical and with low frequency or duration) and other specified ED. The performance of ExpaliTM was evaluated on data from patients referred to the Nutrition Department including a precise DSM-5 diagnosis of ED, a positive SCOFF test (at least 2 "yes" answers) and BMI. Sensitivity, specificity values with a 95% confidence interval (95% CI) and Youden index were calculated for each category.

ELIGIBILITY:
Inclusion Criteria:

* eating disorders
* SCOFF test = 2 or more

Exclusion Criteria:

* no eating disorders
* SCOFF test = 0 or 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited in the Nutrition Department of Rouen University Hospital (France) for suspicion of Eating disorders
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Sensivity and specificity of the clinical algorithm | inclusion